CLINICAL TRIAL: NCT06801392
Title: The Acute Efficacy and Safety of Left Atrial Posterior Wall and Mitral Isthmus Ablation in Patients With Non-Paroxysmal Atrial Fibrillation
Brief Title: Left Atrial Posterior Wall and Mitral Isthmus PF Ablation in Non-Paroxysmal AF Patients
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Varipulse_efficacy_and_safety
Record Dates: First submitted 2025-01-10; First posted 2025-01-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; pulsed-field ablation; varipulse
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ablation strategy 1: PVI + three pairs of overlapping lesions on the posterior wall, mitral isthmus ablation optional
  Interventions: Procedure: pulsed-field ablation
- Ablation strategy 2: PVI + three single lesions on the posterior wall, mitral isthmus ablation optional
  Interventions: Procedure: pulsed-field ablation
- Ablation strategy 3: PVI + four single lesions on the posterior wall, mitral isthmus ablation optional
  Interventions: Procedure: pulsed-field ablation
- Ablation strategy 4: PVI + four pairs of overlapping lesions on the posterior wall, mitral isthmus ablation optional
  Interventions: Procedure: pulsed-field ablation

INTERVENTIONS:
Procedure: pulsed-field ablation — PVI + PW ablation

SUMMARY:
An observational study evaluating efficacy and safety of the Varipulse catheter in pulsed-field ablation of atrial fibrillation

DETAILED DESCRIPTION:
Background: Pulmonary vein (PV) isolation (PVI) is the cornerstone of catheter-based treatment of atrial fibrillation (AF). The left atrial posterior wall (LAPW) and mitral isthmus (MI) are potential ablation targets in patients with non- paroxysmal atrial fibrillation. The efficacy of PVI, LAPW, and MI ablations in early studies of pulse field ablation (PFA) using pentaspline PFA catheters (Farawave, BSCI) or, recently, PVI using a variable-loop circular catheter (Varipulse, Biosense) have been excellent. Complete PV isolation was achieved after first-pass ablation in almost 100% of PVs. Concerning the Farawave catheter, the majority of centers perform empiric pulsed-field PVI, using standard recommended configurations and power settings for ablation catheters, but without verifying PVI (or other lesion using a standard Lasso catheter for and voltage and activation mapping). The praxis regarding LAPW and MI ablations differs significantly among centers; while some centers routinely verify mitral isthmus block using a CS catheter and stimulation maneuvers, others perform anatomicaly-guided MI ablations without block verification by stimulation maneuvers. The ADVENT trial showed that radiofrequency and PF ablations have similar efficacy. However, several cases of PV, LAPW, and MI reconnections have been reported (either acutely or during redo procedures) after ablations using Farawave ablation catheters. In our experience, the efficacy of first-pass PVI using Farawave ablation PF catheters is ~96% (when PV-isolation was verified using a standard Lasso catheter after ablation, data under review). In comparison, first-pass MI block is about ~ 60% (verified using pacing from the left atrial appendage, data under review). Regarding the Varipulse catheter, which recently received the CE mark, efficacy data on PV, LAPW, and MI ablations remains scarce. This raises the question of whether anatomicaly- guided LA ablations (i.e., fluoroscopy and ICA navigation with the recommended ablation setup) should be considered less desirable than LA ablations in which PVI, LAPW, and MI block are verified with additional mapping. With regard to LAPW ablation, the results with pulsed-filed ablation are excellent, and LAWP was isolated in the majority of cases. On the other hand, regarding MI block and based on our previous experience with MI ablations, the probability that a complete block is achieved based solely on an empiric ablation (without verification using either differential pacing, or optimally using 3D mapping) is not high. The advent of the Varipulse system allows for high-power ablations using PF energy combined with 3D mapping capability. As such, it presents a unique opportunity to verify ablation lesions, i.e., verifying the completeness of PVI, LAPW and MI block and locating the most common sites of gaps. Information about the success rate of Varipulse in achieving a complete first-pass LAPW isolation, and MI block, and potentially identifying gaps in the LAPW or in the absence of a MI block could increase first-pass ablation success rates. Regarding LAPW, since an excessive number of PF application could lead to extensive hemolysis or even to worsening of renal function (see below), information about the minimum number of PF energy applications that will already be associated with complete LAPW isolation (complete line between right and left PVs) is of importance. After an initial excellent safety profile for PFA, as more experience was gained with the method, some potential renal issues associated with PFA began to appeared. Recently, a case of renal failure due to hemolysis after PFA using a Farapulse was described. All cases of renal failure occurred after a large number (more than 120) of PF applications using the Farapulse system. The hemolysis is present during pulsed-field ablation, and as our and also other recent data indicates, the amount of hemolysis correlates with the number of PF applications (using Farapulse system). In the study conducted by the investigators, the concentration of red blood cell microparticles (i.e., fragments of destroyed erythrocytes) and other markers hemolysis (e.g. lactate dehydrogenase) correlated with the number of PF applications using Farapulse system. Since the information on hemolysis is new, the "safe" threshold, i.e. the safe number of PF energy application has been still not established. Moreover, since the impulse characteristics differ between different PF systems, it is unclear whether our Farapulse system data can be easily transferred to other PF generators with different pulse characteristics. Determining the amount of hemolysis, renal function and activation of platelets and coagulation after PF ablations using a Varipulse system is the second (safety) part of this project.

Objective: (1) to assess the efficacy of ablation of LAPW and to determine the location of typical gaps after LAPW, (2) to assess the efficacy of ablation of MI and to determine the location of typical gaps after MI, (3) to assess hemolysis during Varipulse ablations, and (4) to analyze activation of thrombotis during Varipulse ablation

Methods: Fifty patients with non-paroxysmal AF will be enrolled. Inclusion criteria will be:

1. non-paroxysmal atrial fibrillation,
2. an indication for catheter ablation according current guidelines,
3. willingness to sign informed content.

Exclusion criteria will be hematological disorders that can be associated with spontaneous hemolysis, chronic kidney disease stage 3 or worse, previous left atrial ablation (either using pulsed-field or radiofrequency energy), conditions associated with increased inflammation (COPD III or more, vasculitis etc.).

The procedure will be performed using fluoroscopy and ICE navigation, analgosedation or general anesthesia will be guided by anesthesiologist. A 10-pole catheter will be placed in the coronary sinus (CS) of all patients. PVI will be performed according to the manufacturer's recommendation similar to how it was done in the inspIRE study (at least 12 applications of PF energy per PV with slight rotation). (2) LAPW ablation will be randomly done in three different settings. The randomization will be stratified according to the LA size.

The ablation settings for LAPW will be following:

1. three pairs of overlapping lesions on the posterior wall (20 patients),
2. three single lesions on the posterior wall (10 patients),
3. four single lesions on the posterior wall (10 patients), and
4. four pairs of overlapping lesions on the posterior wall (10 patients).

The MI will be optional, and MI will be ablated based on the position of the transseptal puncture and the operator's preference, either posteriorly (between the LIPV and the MI annuls) or anteriorly (between the base of the LAA and the MI annulus), and at least three pairs of lesions (with small movement of catheter between each pair) will be applied.

Immediately after the last application of PE energy, and after a 20-minute wait, all lesions will be verified by careful 3D-electro-anatomical mapping (voltage and activation mapping) using Varipulse catheter. Gaps will be located and closed, and the locations of frequent gaps (PVI, LAPW, MI) will be collected. 3D mapping will be repeated in patients with secondarily closed gaps after an additional 20-minute waiting period. All patients will receive additional 1000 mL fluids (saline infusion) immediately after the procedure as kidney protection.

Blood samples will be taken

1. at the beginning of the procedure from the femoral vein,
2. at the end of all ablations before sheath removal, and (3) in the morning on the day after the procedure.

Markers of hemolysis, renal function, and thrombosis. With regard to the hemolytic markers, the concentration of red blood cell microparticles (using flow cytometry) and lactate dehydrogenase will be determined. Furthermore, in relation to hemolysis, renal function (assessed using serum creatinine, and neutrophil gelatinase-associated lipocalin (NGAL) will be determined one day after ablation and compared to baseline values. With regard to the markers of thrombosis, platelet activation markers (CD62P, CD42b and PAC-1), prothrombin fragments and platelet-thrombotic microparticles will be determined.

All adverse event (stroke, pericardial effusion, clinical-apparent coronary spasm, cardiac tamponade) will be evaluated as it is obvious in studies on catheter ablation.

Conclusion: The study will show the efficacy of the ablation (and different number of PF applications) of posterior wall and mitral isthmus using a Varipulse catheter. Data regarding efficacy the location of frequent MI ablation gaps collected during our study should also significantly improve ablation protocols. Finally, the study will assess if PFA using Varipulse is associated with hemolysis, worsening renal function, or activation of thrombotic markers.

ELIGIBILITY:
Inclusion Criteria:

1. non-paroxysmal atrial fibrillation
2. an indication for catheter ablation according current guidelines
3. willingness to sign informed content.

Exclusion Criteria:

1. hematological disorders that can be associated with spontaneous hemolysis
2. chronic kidney disease stage 3 or worse
3. previous left atrial ablation (either using pulsed-field or radiofrequency energy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AF ablation indication
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Acute Success of the Left Atrial Posterior Wall Ablation | during the procedure
  After the last application of PE energy, and after a 20-minute wait, all lesions will be verified by careful 3D-electro-anatomical mapping (voltage and activation mapping) and by conventional pacing manoeuvres.
Acute Success of the Mitral Isthmus Ablation | during the procedure
  After the last application of PE energy, and after a 20-minute wait, all lesions will be verified by careful 3D-electro-anatomical mapping (voltage and activation mapping) and by conventional pacing manoeuvres.
Serum Creatinine Concentration | Blood samples will be taken (1) at the beginning of the procedure from the femoral vein and (2) in the morning on the day after the procedure.
  Serum creatinine concentration
Serum Cystatin C Concentration | Blood samples will be taken (1) at the beginning of the procedure from the femoral vein and (2) in the morning on the day after the procedure.
  Serum cystatin C concentration.
Serum Neutrophil Gelatinase-Associated Lipocalin Concentration | Blood samples will be taken (1) at the beginning of the procedure from the femoral vein and (2) in the morning on the day after the procedure.
  Serum neutrophil gelatinase-associated lipocalin (NGAL).
Red Blood Cell Microparticles | Blood samples will be taken (1) at the beginning of the procedure from the femoral vein, (2) at the end of all ablations before sheath removal, and (3) in the morning on the day after the procedure.
  The concentration of red blood cell microparticles (using flow cytometry).
Lactate Dehydrogenase | Blood samples will be taken (1) at the beginning of the procedure from the femoral vein, (2) at the end of all ablations before sheath removal, and (3) in the morning on the day after the procedure.
  Serum lactate dehydrogenase will be determined.
Platelet Activation Markers | Blood samples will be taken (1) at the beginning of the procedure from the femoral vein, (2) at the end of all ablations before sheath removal, and (3) in the morning on the day after the procedure.
  The platelet activation markers (CD62P, CD42b and PAC-1) will be determined
Prothrombosis Fragments | Blood samples will be taken (1) at the beginning of the procedure from the femoral vein, (2) at the end of all ablations before sheath removal, and (3) in the morning on the day after the procedure.
  Prothrombin fragments will be determined
Platelet-Thrombotic Microparticles | Blood samples will be taken (1) at the beginning of the procedure from the femoral vein, (2) at the end of all ablations before sheath removal, and (3) in the morning on the day after the procedure.
  Platelet-thrombotic microparticles will be determined

OTHER OUTCOMES:
Procedure complications assessment | 0 - 30 days after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided